CLINICAL TRIAL: NCT01884883
Title: Evaluation of a Distraction-rotation Knee Unloader Brace in Patients With Medial Knee Osteoarthritis.
Acronym: ORFEVRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAILLEFERT 2010
Record Dates: First submitted 2013-06-18; First posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

ARMS (1):
- Internal unicompartmental knee brace (Other)
  Interventions: Device: PROTEOR Internal unicompartmental knee brace

INTERVENTIONS:
Device: PROTEOR Internal unicompartmental knee brace
  Other Names: trademark : " PROTEOR " : code name 2H-200

SUMMARY:
The aim of this study is to confirm the biomechanical effects and evaluate functional benefits of a new knee brace combining valgus inducing effect on medial compartment and leg external rotation during the stance phase in patients with symptomatic medial knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient understanding simple order and able to give written consent.
* Man or woman with age between 40 et 75 years
* Unilateral medial symptomatic knee osteoarthritis, defined using the American College of Rheumatology classification
* Radiologic grade II, III ou IV (Kellgren et Lawrence (KL) classification)
* Medial knee compartment (Medial K&L g rade higher than lateral K&L grade
* Knee pain > 40/100 on visual analog scale and <30/100 for the other
* No change in medical treatment for at least 3 months.
* Latest radiographic image < 12 months before inclusion

Exclusion Criteria:

* Patient without healthcare insurance.
* Inflammatory knee arthritis,
* Indication of knee surgery
* Pregnancy, breastfeeding
* Associate neurologic or orthopaedic affection that interferes with gait analysis
* Rapidly destructive arthritis.
* Alzheimer's disease, Parkinson's disease, motor neuronal disorders
* Patient under guardianship or tutelage

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pain score on visual analogic scale | Baseline
  Pain was self-evaluated by patient on visual analogic scale (VAS: 0-100, 0 = no pain at all; 100 = worst pain appendix 1). Such pain is widely used and validated in the literature for the evaluation of knee osteoarthritis treatment outcome.
Pain score on visual analogic scale | Baseline + 5 weeks
  Pain was self-evaluated by patient on visual analogic scale (VAS: 0-100, 0 = no pain at all; 100 = worst pain appendix 1). Such pain is widely used and validated in the literature for the evaluation of knee osteoarthritis treatment outcome.

SECONDARY OUTCOMES:
Evaluation of the functional capacities: KOOS questionnaire. | baseline
Evaluation of the functional capacities: KOOS questionnaire. | baseline + 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francis Maillefert, Principal Investigator — CHU Dijon - Department of Rheumatology
Locations (1):
- CHU de Dijon, Dijon, France